CLINICAL TRIAL: NCT03571594
Title: A Randomized, Double-blind, Placebo-Controlled, Four- Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-5788 in Healthy Adult Volunteers
Brief Title: A Four-Part Study to Assess the Safety, Tolerability, PK and PD of ONO-5788 in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study met a pre-defined protocol study stopping criteria
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-5788-01
Record Dates: First submitted 2018-06-01; First posted 2018-06-27 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind (Parts A, B &C). Open-label (Part D only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- ONO-5788 Part A1 (Experimental): Single ascending doses of ONO-5788 or placebo in fasted healthy volunteers randomized 6 active : 2 placebo per group
  Interventions: Drug: ONO-5788
- ONO-5788 Placebo Part A1 (Placebo Comparator): Single ascending doses of ONO-5788 or placebo in fasted healthy volunteers randomized 6 active : 2 placebo per group
  Interventions: Drug: ONO-5788 Placebo
- ONO-5788 Part A2 (Experimental): Single dose (1-2 groups) of ONO-5788 or placebo in healthy volunteers under fed conditions randomized 6 active : 2 placebo per group
  Interventions: Drug: ONO-5788
- ONO-5788 Placebo Part A2 (Placebo Comparator): Single dose (1-2 groups) of ONO-5788 or placebo in healthy volunteers under fed conditions randomized 6 active : 2 placebo per group
  Interventions: Drug: ONO-5788 Placebo
- ONO-5788 Part B (Experimental): Multiple ascending doses of ONO-5788 or placebo in healthy volunteers randomized 8 active : 2 placebo per group
  Interventions: Drug: ONO-5788
- ONO-5788 Placebo Part B (Placebo Comparator): Multiple ascending doses of ONO-5788 or placebo in healthy volunteers randomized 8 active : 2 placebo per group
  Interventions: Drug: ONO-5788 Placebo
- ONO-5788 Part C (Experimental): Single doses of ONO-5788 or placebo in elderly female or elderly male healthy volunteers randomized 6 active : 2 placebo per group
  Interventions: Drug: ONO-5788
- ONO-5788 Placebo Part C (Placebo Comparator): Single doses of ONO-5788 or placebo in elderly female or elderly male healthy volunteers randomized 6 active : 2 placebo per group
  Interventions: Drug: ONO-5788 Placebo
- ONO-5788 Part D (Experimental): Single doses of ONO-5788, octreotide or placebo in healthy volunteers stimulated with growth hormone release hormone (GHRH) and arginine
  Interventions: Drug: ONO-5788
- ONO-5788 Placebo Part D (Placebo Comparator): Single doses of ONO-5788, octreotide or placebo in healthy volunteers stimulated with growth hormone release hormone (GHRH) and arginine
  Interventions: Drug: ONO-5788 Placebo
- Octreotide Part D (Active Comparator): Single doses of ONO-5788, octreotide or placebo in healthy volunteers stimulated with growth hormone release hormone (GHRH) and arginine
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: ONO-5788 — Investigational drug
  Arms: ONO-5788 Part A1; ONO-5788 Part A2; ONO-5788 Part B; ONO-5788 Part C; ONO-5788 Part D
Drug: ONO-5788 Placebo — Placebo Comparator
  Arms: ONO-5788 Placebo Part A1; ONO-5788 Placebo Part A2; ONO-5788 Placebo Part B; ONO-5788 Placebo Part C; ONO-5788 Placebo Part D
Drug: Octreotide — Active Comparator in Part D
  Other Names: Sandostatin
  Arms: Octreotide Part D

SUMMARY:
This is a first in human study to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of ONO-5788 in healthy adult volunteers. This study will be conducted in 4 parts: a single-ascending dose part, a multiple-ascending dose part, an elderly part and a proof of principle part.

DETAILED DESCRIPTION:
This single centre study will be comprised of 4 parts, Part A (SAD; up to 7 cohorts, 8 subjects per cohort and including an assessment of food effect), a multiple-dose part (up to 4 doses, 10 subjects per cohort); an elderly cohort (8 subjects per gender) and a proof of principle part.

The single ascending dose part (Part A) comprises of increasing doses of an oral solution or capsule, with an investigation of the potential for food effects.

The multiple ascending dose part (Part B, MAD; 14 days dosing) will be initiated after the PK and safety data are available from the single ascending dose part. Subjects in Part B will have ultrasound scans of the gallbladder during the study and at screening a HIDA scan will be performed. An evaluation of the PK in the elderly and any potential gender differences will also be evaluated in Part C. Subjects in Part C will have an ultrasound of the gallbladder at screening.

Part D will be a proof of principle evaluation where the effects of ONO-5788 to inhibit the GHRH and arginine-stimulated GH release will be evaluated. Octreotide acetate is a reference arm in this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male and female (women of non-child bearing potential, surgically sterile) volunteers, 18-55 years of age, inclusive, at screening (Parts A & B only).
* Healthy, adult, males and female (women of non-child bearing potential), ≥65 years of age at screening (Part C only).
* Healthy, adult, male, 18-40 years of age, inclusive, at screening (Part D only).
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECG abnormalities (All Parts).
* Body mass index (BMI) of ≥18.5 to ≤30 kg/m2 at screening (Parts A, B & C).
* Body mass index (BMI) of ≥18.5 to <25 kg/m2 at screening (Part D only).

Exclusion Criteria:

* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs,excipients or related compounds.
* History or presence of:

  1. Gallstones, cholangitis, and/or cholecystitis or clinically significant findings on gallbladder ultrasound as determined by the Principal Investigator;
  2. Pancreatitis;
  3. Hypothyroidism;
  4. Known diabetes mellitus type 1 or type 2;
  5. Hypocalcaemia or hypokalemia;
  6. Hypoglycemia or hyperglycemia or fasting blood glucose outside normal local range;
  7. Thrombocytopenia or other clinically significant hematologic abnormalities;
  8. Inflammatory bowel disease, irritable bowel syndrome, or abdominal surgery;
  9. Known vitamin B12 deficiency.
  10. Abnormal gallbladder ejection fraction on hepatobiliary iminodiacetic acid (HIDA) scan at screening (Part B only)
* Positive urine drug, alcohol or cotinine results at screening or check in.
* Clinically significant serum electrolyte (sodium, potassium, chloride, bicarbonate) abnormalities at screening or each check-in, in the estimation and clinical judgment of the PI or designee.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Seated blood pressure is less than 90/40 millimeter of mercury (mmHg) or greater than 140/90 mmHg (160/95 mmHg for Part C) at screening.
* Has engaged in strenuous physical exercise in the 48 hours prior first dosing or intends to undergo strenuous physical exercise at any time throughout the study.
* Donation of blood or significant blood loss within 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For parts A and B male and females of non-childbearing potential will be recruited. For part C both elderly males and elderly females (of non-childbearing potential) will be recruited. For Part D only males will be recruited.
Enrollment: 76 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events by severity | Part A - up to day 8; Part B - at least day 21; Part C - at least day 21; and Part D - up to day 28
  An adverse event is any untoward medical occurrence in a participant who receive study drug without regard to possible causal relationship.
Number of participants with serious adverse events (SAEs) | Part A - up to day 8; Part B - at least day 21; Part C - at least day 21; and Part D - up to day 28
  An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged hospitalization, life-threatening experience or persistent disability.
Number of participants with clinically significant changes in vital signs | Part A - up to day 8; Part B - at least day 21; Part C - at least day 21; and Part D - up to day 28
  Number of participants with clinically significant changes in vital signs including pulse/heart rate, respiratory rate, and blood pressure will be reported.
Number of participants with ECG abnormalities | Part A - up to day 8; Part B - at least day 21; Part C - at least day 21; and Part D - up to day 28
  Number of participants with ECG abnormalities will be reported
Number of participants with clinical laboratory abnormalities | Part A - up to day 8; Part B - at least day 21; Part C - at least day 21; and Part D - up to day 28
  Number of participants with clinical laboratory abnormalities will be reported
Number of participants with clinically significant change in ultrasound of gallbladder | Part B - up to day 21
  Number of participants with clinically significant change in ultrasound of gallbladder will be reported

SECONDARY OUTCOMES:
Pharmacokinetics (AUC) | Day 1 through Day 14
  Assessment of the plasma area under the curve of ONO-5788 and metabolites (Parts A, B and C only)
Pharmacokinetics (AUC) - food effect | Day 1
  Effect of food on the plasma area under the curve of ONO-5788 and metabolites (Parts A only)
Pharmacokinetics (Cmax) | Day 1 through Day 14
  Assessment of the maximum observed plasma concentration of ONO-5788, metabolites (Parts A, B, C & D) and octreotide (Part D only)
Pharmacokinetics (Cmax) - food effect | Day 1
  Effect of food on the maximum observed plasma concentration of ONO-5788, and metabolites (Part A only)
Pharmacokinetics (Tmax) | Day 1 through Day 14
  Assessment of the time to reach Cmax for ONO-5788, metabolites (Parts A, B, C & D) and octreotide (Part D only)
Pharmacokinetics (Tmax) - food effect | Day 1 through Day 14
  Effect of food on the time to reach Cmax for ONO-5788, metabolites (Part A only)
Pharmacokinetics (Ctrough) | Day 1 through Day 14
  Assessment of trough levels for ONO-5788 and metabolites immediately before dosing (Part B only)
Pharmacokinetics (T1/2) | Day 1 through Day 14
  Assessment of the elimination half-life of ONO-5788 and metabolites (Parts A, B and C only)
Pharmacokinetics (T1/2) - food effect | Day 1
  Effect of food on the elimination half-life of ONO-5788 and metabolites (metabolite) (Part A only)
Pharmacokinetics (CL/F) | Day 1
  Assessment of the apparent clearance rate of ONO-5788 (Parts A & C)
Pharmacokinetics (CL/F) - food effect | Day 1
  Effect of food on the apparent clearance rate of ONO-5788 (Part A only)
Pharmacokinetics (Cave) | Day 1
  Average concentration of ONO-5788/metabolites/Octreotide (Part D only)
Pharmacodynamics (IGF-1) | Day 1 through Day 21
  Assessment of the effects of ONO-5788 on IGF-1 levels (Part B only)
Pharmacodynamics (Growth Hormone) | Day 1 through Day 21
  Assessment of the effects of ONO-5788 on GH levels (Part B)
Pharmacodynamics (Growth Hormone) | Day 1
  Assessment of the effects of ONO-5788 on GHRH & arginine stimulated GH levels (Part D)
Pharmacodynamics (IGFBP3) | Day 1 through Day 21
  Assessment of the effects of ONO-5788 on IGFBP3 levels (Part B only)

CONTACTS AND LOCATIONS:
Overall Officials: Terry O'Reilly, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States